CLINICAL TRIAL: NCT00783510
Title: A Long-term, Multi-center, Longitudinal Post-marketing, Observational Study to Assess Long Term Safety and Effectiveness of HUMIRA® (Adalimumab) in Children With Moderately to Severely Active Polyarticular or Polyarticular-course Juvenile Idiopathic Arthritis (JIA) - STRIVE
Brief Title: Juvenile Idiopathic Arthritis (JIA) Registry
Acronym: STRIVE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P10-262
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Juvenile Idiopathic Arthritis; JIA
Keywords: JIA; Juvenile Idiopathic Arthritis; Juvenile Arthritis; Polyarticular JIA; Polyarticular-course JIA
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HUMIRA® Treatment Arm: For patients taking HUMIRA®
  Interventions: Biological: adalimumab
- Methotrexate Treatment Arm: For patients taking Methotrexate
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Biological: adalimumab — As prescribed by treating physician
  Other Names: HUMIRA®
  Groups: HUMIRA® Treatment Arm
Drug: Methotrexate — As prescribed by treating physician
  Other Names: MTX
  Groups: Methotrexate Treatment Arm

SUMMARY:
This is a global registry, to evaluate the long-term safety of Humira® in patients with moderate to severe polyarticular Juvenile Idiopathic Arthritis (JIA), that are treated as recommended in the Humira® product label. Patients treated with MTX will be considered a reference group. Patients will be followed in both the Humira® and Methotrexate (MTX) arms for 10 years from the enrollment date into one of the treatment arms.

DETAILED DESCRIPTION:
This registry will assess the incidence and rate of Humira (monotherapy or combination therapy with MTX) or MTX observational and treatment-emergent SAEs, Adverse Events of Special Interest (AESI) and Pregnancy in patients diagnosed with moderately to severely active polyarticular or polyarticular-course JIA through Year 5. From Year 6 through Year 10 SAEs, a subset of AESI that includes congestive heart failure (CHF), malignancies, AEs at least possibly related to and/or leading to discontinuation of registry treatment and pregnancies will be collected. For JIA patients 2 to< 4 years of age in countries with available local approval for this group of patients at the time of consent to the registry, emergent AESI, SAEs and pregnancy (at the age when a patient can become pregnant) will be collected for the full 10 years. The approved age range for HUMIRA in the U.S., European Union (EU) and in Australia is 4 years of age and older, and recent approval in EU for JIA patients 2 to < 4 years of age.

Patients who discontinue from the registry before 10 years will be offered to participate in the direct to Health Care Provider follow-up process, as allowed by local regulations.

ELIGIBILITY:
Inclusion Criteria:

* For a patient enrolling into the HUMIRA® arm; a pediatric patient diagnosed at any time with moderately to severely active polyarticular or polyarticular-course JIA (defined as arthritis affecting >= 5 joints at the time of diagnosis of polyarticular or polyarticular-course JIA) who has been prescribed HUMIRA® therapy according to the local approved HUMIRA® product labeling and meets one of the following criteria:
* Enrolled patients are 4 to 17 years of age as per approved HUMIRA® product label with the addition of JIA patients 2 to < 4 years of age in countries with available local approval for this group of patients at the time of consent to the registry.
* Newly initiated (within 24 months of registry entry) on HUMIRA® therapy and has received continuous (no more than 70 consecutive days off drug) HUMIRA® therapy, and the physician can provide available source documentation of SAEs, AEs of Special Interest, and dosing information since initiation of therapy;
* Or is entering after participation (within 24 months of registry entry or, if longer, continuously treated at the same site) in an AbbVie Humira sponsored study, regardless of age or the number of joints with symptoms of JIA, and has received continuous (no more than 70 consecutive days off drug) HUMIRA® therapy and the physician can provide available source documentation of SAEs, AEs of Special Interest, and dosing information since initiation of therapy.
* For a patient enrolling into the MTX arm; a pediatric patient diagnosed at any time with moderately to severely active polyarticular or polyarticular-course JIA (defined as arthritis affecting >= 5 joints at the time of diagnosis of polyarticular or polyarticular-course JIA) who is prescribed MTX therapy alone or in combination with other disease modifying anti-rheumatic drugs (DMARDs) according to the local product labeling (initiated treatment within 24 months of registry entry) and has received continuous therapy and the physician can available provide source documentation of SAEs, AEs of Special Interest, and dosing information since initiation of therapy.
* Patients who were treated in the MTX arm of this registry and prematurely discontinued from the MTX arm due to being a non-responder, or became intolerant of MTX treatment or are in need of combination treatment with HUMIRA® therapy may be eligible to enroll into the HUMIRA® treatment arm if all ongoing AEs/SAEs have been resolved, and they meet inclusion criteria and can enroll within the registry enrollment period. In case of ongoing AEs/SAEs at the time of the treatment arm switch, the AbbVie Designated Physician should be contacted to assess the eligibility of patient to roll into Humira treatment arm.
* Parent or guardian has voluntarily signed and dated an informed consent/patient authorization form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) if applicable according to local law, after the nature of the registry has been explained and the patient's parent or legal guardian has had the opportunity to ask questions. Pediatric patients will be included in all discussions as per applicable local regulations in order to obtain verbal or written assent.

Exclusion Criteria:

* Patients should not be enrolled into the HUMIRA® or Methotrexate (MTX) arm if they cannot be prescribed and treated in accordance with the approved local HUMIRA® and/or with the local MTX product label
* Patients should not be enrolled into the HUMIRA® or MTX arm if they require on-going treatment with Kineret® (anakinra), Orencia® (abatacept), Rituxan® (rituximab), Enbrel® (etanercept), and Remicade® (infliximab), or any other approved biologic agents or investigational agents.
* Patients should not be enrolled into the MTX arm if they have had prior treatment with any investigational agent or anti-rheumatic biologic therapy such as, but not limited to, Orencia® (abatacept), Enbrel® (etanercept), Remicade® (infliximab), Rituxan® (rituximab), or Actemra® (tocilizumab)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who are diagnosed at any time with moderately to severely active polyarticular or polyarticular-course JIA, (defined as arthritis affecting greater than 5 joints at the time of diagnosis of polyarticular or polyarticular-course JIA), prescribed and treated in a routine clinical setting either with Humira® (adalimumab), or MTX. Approximately 800 patients will be enrolled in the United States, EU countries, and Australia. Approximately 40 to 45 physicians will be included based on participation in prior AbbVie Humira sponsored clinical JIA studies.
Sampling Method: Non-Probability Sample
Enrollment: 849 (Actual)
Dates: Start 2008-07-11 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events (SAEs) | Up to 10 years
  Collected as events occur during the registry and as part of prior clinical studies. Events are collected retrospectively for patients who dosed prior to enrollment in the registry and as part of the Health Care Provider (HCP) process.
Incidence of Adverse Events (AEs) of Interest | Up to 10 years
  Collected as events occur during the registry and as part of prior clinical studies. Events are collected retrospectively for patients who dosed prior to enrollment in the registry and as part of the Health Care Provider (HCP) process.

SECONDARY OUTCOMES:
Pediatric American College of Rheumatology (PedACR) 50 | Up to 10 years
  Effectiveness data will be analyzed as observed and will be summarized for All Treated Patient Population.
Pediatric American College of Rheumatology (PedACR) 70 | Up to 10 years
  Effectiveness data will be analyzed as observed and will be summarized for All Treated Patient Population.
Pediatric American College of Rheumatology (PedACR) - 30 | Up to 10 years
  Effectiveness data will be analyzed as observed and will be summarized for All the Treated Patient Population.
Child Health Questionnaire (CHQ-PF50) | Assessed in months 1,3, 6 and every 6 months through Year 5
  The results will be summarized at each visit and will be used in exploratory analyses.
Pediatric American College of Rheumatology (PedACR) 90 | Up to 10 years
  Effectiveness data will be analyzed as observed and will be summarized for All Treated Patient Population.
Juvenile arthritis disease activity score (JADAS) | Assessed in months 1,3, 6 and every 6 months through Year 5
  Effectiveness data will be analyzed as observed and will be summarized for All Treated Patient Population. Is the total scores of four activity scales (Physician's Global Assessment of patient's disease, Parents' Global Assessment of patient's overall well-being, Number of active joints and Normalized erythrocyte sedimentation rate (ESR) if collected and available.
Physical function of the Disability Index of Childhood Health Assessment Questionnaire (DIHAQ) | Assessed in months 1,3, 6 and every 6 months through Year 5
  Effectiveness of therapy through clinical assessment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (92):
- United States (32):
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 21023, Phoenix, Arizona
  - Catalina Pointe Clinical Research /ID# 40227, Tucson, Arizona
  - Arkansas Children's Hospital /ID# 23505, Little Rock, Arkansas
  - Children's Hospital Los Angeles /ID# 24386, Los Angeles, California
  - Children's National Medical Center /ID# 23506, Washington D.C., District of Columbia
  - Duplicate_Arthritis Associates South FL /ID# 17001, Delray Beach, Florida
  - Ann & Robert H Lurie Children's Hospital of Chicago /ID# 20966, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 21981, Chicago, Illinois
  - Methodist Medical Group Rheum /ID# 46343, Peoria, Illinois
  - Indiana University /ID# 11421, Indianapolis, Indiana
  - University of Louisville /ID# 23507, Louisville, Kentucky
  - Arthritis Care Spec. of MD /ID# 21961, Ellicott City, Maryland
  - Tufts Medical Center /ID# 21965, Boston, Massachusetts
  - Creighton Univ Med Ctr /ID# 11423, Omaha, Nebraska
  - St. Barnabas Ambulatory Care /ID# 21025, West Orange, New Jersey
  - North Shore University Hospital /ID# 21022, New Hyde Park, New York
  - University of Rochester Medical Center /ID# 20967, Rochester, New York
  - New York Medical College /ID# 21964, Valhalla, New York
  - Duke Cancer Center /ID# 22904, Durham, North Carolina
  - Bone Spine Sports/Medctr One /ID# 21962, Bismarck, North Dakota
  - Akron Children's Hospital /ID# 22907, Akron, Ohio
  - University of Cincinnati /ID# 14101, Cincinnati, Ohio
  - Nationwide Children's Hospital /ID# 21963, Columbus, Ohio
  - Legacy Emanuel Medical Center /ID# 14102, Portland, Oregon
  - St. Christopher's Hospital /ID# 24385, Philadelphia, Pennsylvania
  - Arthritis Associates of Kingsport /ID# 44462, Kingsport, Tennessee
  - Dr. Ramesh Gupta /ID# 45342, Memphis, Tennessee
  - Scott & White Health Care /ID# 36762, Round Rock, Texas
  - University of Utah /ID# 21041, Salt Lake City, Utah
  - Children's Speciality Center /ID# 11503, Burlington, Vermont
  - Seattle Children's Hospital /ID# 20968, Seattle, Washington
  - Children's Hospital Wisconsin - Milwaukee Campus /ID# 40226, Milwaukee, Wisconsin
- Duplicate_Womens and Childrens Hospital /ID# 59182, Adelaide, South Australia, Australia
- Austria (4):
  - Medizinische Universitaet Graz /ID# 26126, Graz, Styria
  - Duplicate_Kepler Universitaetsklinikum GmbH /ID# 39068, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 26127, Vienna, Vienna
  - Landeskrankenhaus Bregenz /ID# 26128, Bregenz, Vorarlberg
- Czechia (4):
  - Fakultni Nemocnice Brno /ID# 37343, Brno
  - Revmatologicky ustav v Praze /ID# 43344, Prague
  - Vseobecna fakultni nemocnice v Praze /ID# 47401, Prague
  - Fakultni Nemocnice v Motole /ID# 37342, Prague
- Denmark (2):
  - Aarhus University Hospital /ID# 25445, Aarhus N, Central Jutland
  - Duplicate_Rigshospitalet, Finsen Centre /ID# 25444, Copenhagen
- France (10):
  - CHU Strasbourg - Hopital de Hautepierre /ID# 25450, Strasbourg, Bas-Rhin
  - Duplicate_CHU Bordeaux - Hopital Pellegrin /ID# 25454, Bordeaux, Gironde
  - CHRU Tours - Hopital Bretonneau /ID# 27126, Tours, Indre-et-Loire
  - CHRU Nancy - Hopitaux de Brabois /ID# 25452, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille - Hopital Claude Huriez /ID# 25449, Lille, Nord
  - CHU Toulouse /ID# 37347, Toulouse, Occitanie
  - AP-HP - Hôpital Bicêtre /ID# 25443, Le Kremlin-Bicêtre
  - Duplicate_AP-HP - Hopital Cochin /ID# 37345, Paris
  - AP-HP - Hopital Necker /ID# 25442, Paris
  - Duplicate_CHU de Rennes - Hospital Sud /ID# 27123, Rennes
- Germany (10):
  - Universitaetsklinikum Tuebingen /ID# 39070, Tübingen, Baden-Wurttemberg
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 41623, Berlin
  - Helios Klinikum Berlin-Buch /ID# 37348, Berlin
  - Klinikum Bremen Mitte /ID# 45942, Bremen
  - Klinikum Dortmund gGmbH /ID# 44003, Dortmund
  - Center Rheumatology Child&Adol /ID# 39069, Garmisch-Patenkirchen
  - Hamburger Zentrum fuer Kinder- und Jugendrheumatologie /ID# 39223, Hamburg
  - Klinikum St. Georg gGmbH /ID# 37349, Leipzig
  - Asklepios Klinik Sankt Augustin /ID# 41622, Sankt Augustin
  - Rheumazentrum Wedel /ID# 37350, Wedel
- Greece (2):
  - Children's Hosp P. A. Kyriakou /ID# 25448, Athens, Attica
  - General Hospital of Thessaloniki Hippokrateio /ID# 25447, Thessaloniki
- Hungary (2):
  - Debreceni Egyetem Klinikai Kozpont /ID# 95863, Debrecen, Hajdú-Bihar
  - Orszagos Reumatologiai es Fizioterapias Intezet /ID# 95095, Budapest
- Italy (10):
  - Azienda Ospedaliero Universitaria Meyer /ID# 26123, Florence, Firenze
  - IRCCS Ospedale Pediatrico Bambino Gesu /ID# 39074, Rome, Roma
  - Duplicate_Azienda Ospedaliera Spedali Civili /ID# 39077, Brescia
  - Duplicate_Universita di Catania /ID# 39075, Catania
  - Ospedale Ss. Annunziata /ID# 37353, Chieti
  - Istituto Giannina Gaslini /ID# 26668, Genova
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 26124, Milan
  - Duplicate_Universita di Napoli Federico II /ID# 39078, Naples
  - Azienda Ospedaliera Universitaria Federico II /ID# 39072, Napoli
  - Fondazione IRCCS Policlinico /ID# 39076, Pavia
- Universitair Medisch Centrum Utrecht /ID# 48842, Utrecht, Netherlands
- Oslo Universitetssykehus, Radiumhospitalet /ID# 46402, Oslo, Norway
- Portugal (3):
  - Hospital Garcia de Orta, EPE /ID# 37355, Almada
  - Centro Hospitalar Universitario de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 42682, Lisbon
  - Centro Hospitalar Universitario do Porto, EPE - Hospital Santo Antonio /ID# 39081, Porto
- Puerto Rico (2):
  - Centro de Reumatologia Pediatrico de Puerto Rico /Id# 61047, Bayamón
  - Puerto Rico Children Hospital /ID# 47742, Bayamón
- Narodny ustav reumatickych chorob /ID# 38102, Piešťany, Slovakia
- Spain (6):
  - Hospital Sant Joan de Deu /ID# 37358, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Severo Ochoa /ID# 41751, Leganés, Madrid
  - Hospital Universitario Vall d'Hebron /ID# 37357, Barcelona
  - Hospital Infantil Universitario Nino Jesus /ID# 37360, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 41624, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 37359, Valencia
- Queen Silvia Children's Hosp /ID# 26125, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P10-262#additional-resources-section